CLINICAL TRIAL: NCT05699629
Title: A Prospective Longitudinal Multi-Omics Cohort of Patients With Coronary Heart Disease Undergoing Coronary Angiography
Brief Title: Prospective Coronary Heart Disease Cohort
Status: Recruiting | Type: Observational
Sponsor: Shandong First Medical University (Other)
Collaborators: Jinan Central Hospital (Other); Shandong Provincial Hospital (Other Government); The Second Affiliated Hospital of Shandong First Medical University (Other); Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-206-02
Record Dates: First submitted 2023-01-09; First posted 2023-01-26 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Coronary Heart Disease; Myocardial Infarction
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and fecal samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the biomarkers for the prognosis of coronary heart disease, patients with coronary heart disease will be recruited and followed up for at least 2 years.

DETAILED DESCRIPTION:
Patients with cardiovascular disease undergoing coronary angiography will be recruited and prospectively followed up for the incidence of major adverse cardiovascular events (MACE events), including all-cause mortality, cardiovascular mortality, ischemic stroke, heart failure and rehospitalization. Blood and fecal samples will be collected for further analysis. The basic and clinical information will be collected such as socio-demographic, diet, lifestyle, psychological status and medical history. The biomarkers for the incidence of coronary heart disease and the factors contributing to the poor prognosis of coronary heart disease will be investigated based on multi-omics analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as coronary heart disease or with unexplained chest pain needed to undergo coronary angiography.
* Healthy subjects undergoing routine physical examination in the physical examination department and willing to sign informed consent will be recruited as control subjects.

Exclusion Criteria:

* With malignant tumors, infectious diseases and advanced liver diseases.
* Won't sign an inform consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with coronary heart diseases undergoing coronary angiography and healthy control subjects undergoing routine physical examination in physical examination department.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2027-01-21 (Estimated); Study Completion 2027-01-21 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events | 2-year outcome and long-term outcome
  all-cause mortality, cardiovascular mortality, ischemic stroke, heart failure and rehospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Tao Xu, Dr., Study Chair — Shandong First Medical University
Locations (1):
- Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No